CLINICAL TRIAL: NCT00741234
Title: A Phase I Dose Escalation Study of Oral SB939 When Administered Thrice Weekly (Every Other Day) for 3 Weeks in a 4-week Cycle in Patients With Advanced Malignancies
Brief Title: A Phase I Dose Escalation Study of Oral SB939 Administered Alone or With Azacitidine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: S*BIO (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SB939-2006-001
Record Dates: First submitted 2008-08-22; First posted 2008-08-26 (Estimated); Last update posted 2012-04-23 (Estimated); Status verified 2012-04

CONDITIONS: Solid Tumors; Hematologic Malignancies; Myelodysplastic Syndrome
Keywords: SB939; Myelodysplastic Syndrome; Combination with azacitidine; Solid malignancies; Hematologic malignancies; HDAC inhibitor; Refractory to standard therapy
MeSH Terms: conditions — Hematologic Neoplasms; Myelodysplastic Syndromes | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): Advanced solid tumors
  Interventions: Drug: SB939
- B (Experimental): Advanced hematologic malignancies
  Interventions: Drug: SB939
- C (Experimental): Myelodysplastic Syndrome
  Interventions: Drug: SB939; Drug: Azacitidine

INTERVENTIONS:
Drug: SB939 — SB939 taken orally in a 4-week cycle.
Drug: Azacitidine — Azacitidine taken orally with SB939 in a 4-week cycle
  Other Names: Vidaza
  Arms: C

SUMMARY:
This is an open label, dose escalation study with 3 arms (Arms A, B, and C). Arm A will assess the safety and tolerability of escalating doses of SB939 in cohorts of patients with advanced solid tumors. Arm B will assess the safety and tolerability of escalating doses in cohorts of patients with advanced hematologic malignancies. Arm C will assess the safety and tolerability of SB939 in combination with standard azacitidine therapy.

ELIGIBILITY:
Inclusion criteria:

Arms A & B:

* Patients with solid tumors in Arm A and hematologic malignancies in Arm B that is classified as intermediate 1 or greater according to the International Prognostic Scoring System (IPSS) risk category for whom therapy is indicated;
* ECOG performance status (PS) 0-2;
* Patients must have adequate non-hematologic organ system function.

Arm C:

* Patients with MDS that is classified as intermediate 1 or greater according to the International Prognostic Scoring System (IPSS) risk category for whom therapy is indicated;
* Have not been treated with azacitidine and are a candidate for treatment with azacitidine;
* ECOG performance status (PS) 0-2;
* Patients must have adequate non-hematologic organ system function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2007-04; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of SB939, administered orally every other day 3 times a week for 3 consecutive weeks, repeated every 4 weeks, either alone (Arms A and B), or in combination with azacitidine therapy in (Arm C). | Throughout the study

SECONDARY OUTCOMES:
To establish the maximum tolerated dose and a recommended phase II dose of SB939 as a single agent when administered every other day 3 times a week for 3 consecutive weeks, repeated every 4 weeks | Throughout the study
To determine the dose limiting toxicities of SB939 | Throughout the study
To determine the pharmacokinetic profile of SB939 | Throughout the study
To assess histone acetylation in PBMC and other biomarkers | Throughout the study
To document anti-tumor activity | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: George Wilding, M.D., Principal Investigator — University of Wisconsin, Madison; Boon Cher Goh, M.D., Principal Investigator — National University Hospital, Singapore; Han Chong Toh, M.D., Principal Investigator — National Cancer Center; Charles Chuah, M.D., Principal Investigator — Singapore General Hospital; Guillermo Garcia-Manero, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (5):
- United States (2):
  - MD Anderson Cancer Center, Houston, Texas
  - University of Wisconsin-Madison, Madison, Wisconsin
- Singapore (3):
  - National University Hospital, Singapore
  - National Cancer Center, Singapore
  - Singapore General Hospital, Singapore